CLINICAL TRIAL: NCT06615219
Title: Effects of Intergroup Contact Training on Aging Stereotypes in Undergraduate Nursing Students: A Randomized Controlled Trial
Brief Title: Intergroup Contact Intervention for Nursing Undergraduates to Improve Aging Stereotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Responsible Party: Principal Investigator, Li Fang, Principal Investigator, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022025.
Record Dates: First submitted 2024-08-27; First posted 2024-09-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Aging; Ageism
MeSH Terms: conditions — Ageism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intergroup contact training + Regular course training (Experimental): In addition to the regular curriculum, the experimental group of nursing students were required to receive the intervention program developed by this study.
  Interventions: Other: Intergroup contact training
- Regular course training only (Active Comparator): Nursing undergraduates in the control group received regular course teaching and practical activities, including geriatric nursing, daily courses and community activities.
  Interventions: Other: Regular course training only

INTERVENTIONS:
Other: Intergroup contact training — The intervention program uses direct contact and four types of indirect contact as the intervention strategy and general framework, and is divided into three main steps, assessing and reflecting on aging stereotypes, carrying out indirect and direct contact, and evaluating the effectiveness of the intervention. The time period is 12 weeks, with the interventionists comprising the researcher and nursing students. The forms of the intervention include holding mini-lectures, organizing participation in voluntary activities, and nostalgia interviews.
  Arms: Intergroup contact training + Regular course training
Other: Regular course training only — The specific process is to sign in the classroom, review the knowledge of the previous class by asking questions, introduce the content of the new class, the teacher explains the knowledge points according to the teaching objectives and teaching content, and finally assigns the post-class homework of the course content. At the end of the experiment, the control group was given compensatory intervention.
  Arms: Regular course training only

SUMMARY:
This study aimed to investigate the effects of intergroup contact training on the levels of aging stereotypes, intergroup anxiety, and willingness to engage in geriatric nursing work among undergraduate nursing students.

DETAILED DESCRIPTION:
This research was designed as a pre-test-post-test randomized controlled experimental study. Nursing students from a university in Hangzhou, China served as the research subjects, who were randomly assigned to the experimental or control group. The control group received training in the regular course and was given compensatory intervention after the experiment, while the experimental group received intergroup contact training (the regular course combined with intergroup contact content). Such training was carried out in the forms of both individual and group interventions for a duration of 12 weeks. The levels of aging stereotypes, intergroup anxiety, and the willingness to engage in geriatric nursing among the nursing students were investigated before and after the training. Number, percentage, mean, standard deviation, Shapiro-Wilk, T-test, Wilcoxon signed ranks tests, and Mann-Whitney U tests were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* full-time undergraduate students enrolled in the nursing program
* not yet enrolled in a geriatric nursing course
* agreed to participate in this study and signed an informed consent form

Exclusion Criteria:

* students in the nursing program pursuing a bachelor degree through a vocational-to-degree pathway
* Students who have taken a break from their studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The implicit effect value (D) | Baseline and Month 3
  The implicit effect value were measured by the Single-Category Implicit Association Test (SC- IAT), a time-limited word categorization task, using the E-Prime procedure. The SC-IAT program consists of four blocks: Blocks I and III are practice blocks, while Blocks II and IV are formal tests. The data analyzed were derived from Blocks II and IV. Blocks I and II feature incompatible tasks with positive words for the elderly on the left and negative words on the right. Blocks III and IV are compatible tasks, with positive words on the right and elderly concept words and negative words on the left. The implicit effect value (D) was calculated by subtracting the mean reaction time of the compatible task from that of the incompatible task, then dividing by the standard deviation of correct reaction times. A D value of 0 indicates a neutral implicit aging stereotype, while a value less than 0 suggests a negtive stereotype.

SECONDARY OUTCOMES:
Geriatric Nursing Willingness Scale | Baseline and Month 3
  The Geriatric Nursing Willingness Scale was used to measure the intention to engage in geriatric nursing. The scale consists of 21 entries divided into four main sections: behavioral attitudes, subjective norms, perceived behavioral control, and behavioral intentions. It was scored on a 5-point Likert scale, with positive entries scoring 10, 8, 6, 4, and 2 in that order, and the reverse for negative entries. The Cronbach' α coefficient in this study was 0.787.
Intergroup Anxiety Scale (IAS) | Baseline and Month 3
  The Intergroup Anxiety Scale was used to measure intergroup anxiety. The scale was developed by Stephan and consists of 10 entries on a 7-point Likert scale. Entries 5 to 7 are reverse scored, with lower scores indicating higher levels of intergroup anxiety. The scale is widely applied internationally, with a Cronbach' α coefficient of 0.808 in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Meijuan Cao, Study Chair — Huzhou University
Locations (1):
- School of Nursing, Hangzhou Normal University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Cao M, Li F, Yao Q, Zhou N, Xiang T, Wu H. Effects of inter-group contact training on aging-related stereotypes among undergraduate nursing students: a randomized controlled trial. Gerontol Geriatr Educ. 2025 Aug 25:1-16. doi: 10.1080/02701960.2025.2551960. Online ahead of print. PMID 40853547